CLINICAL TRIAL: NCT00015444
Title: Screening and Natural History: Primary Lateral Sclerosis and Related Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010145; 01-N-0145
Record Dates: First submitted 2001-04-18; First posted 2001-04-19 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-04-24

CONDITIONS: Primary Lateral Sclerosis
Keywords: Apparently Sporadic Spastic Paraplegia; Spasticity; Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Muscle Stiffness; Involuntary Muscle Contraction; Isaacs Syndrome
MeSH Terms: conditions — Motor Neuron Disease; Muscle Spasticity; Amyotrophic Lateral Sclerosis; Dyskinesias; Isaacs Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Objective:

The objectives of this protocol are:

to develop and maintain a repository of clinically characterized patients with primary lateral sclerosis for future research protocols,

to characterize the natural history of neurodegenerative disorders with corticospinal neuron degeneration,

to investigate proposed etiologies, risk factors, and biomarkers for the development of these disorders and for disease progression

Study Population:

240 patients with adult-onset progressive spasticity with a diagnosis of primary lateral sclerosis or related upper motor neuron disorder

Design:

Patients who have been referred by physicians for primary lateral sclerosis will undergo a screening evaluation at the first visit. The screening visit will include review of outside medical records, neurological examination, and diagnostic testing to determine possible causes of spasticity. Patients fulfilling the clinical criteria for primary lateral sclerosis by history or examination will be followed to determine the natural history of this disorder. Measures of motor and cognitive function will be made at baseline and follow-up visits to follow clinical progression. Magnetic resonance imaging will be carried out to determine if imaging changes occur over time. Patients identified in this protocol who are eligible for other research protocols will be invited to participate in additional protocols.

Outcome Measures:

Clinical progression will be documented by measures of finger-tapping, timed gait, speech. The association between clinical progression and MRI measures will be assessed as a secondary outcome....

DETAILED DESCRIPTION:
Objective:

The objectives of this protocol are:

* to develop and maintain a repository of clinically characterized patients with primary lateral sclerosis for future research protocols,
* to characterize the natural history of neurodegenerative disorders with corticospinal neuron degeneration,
* to investigate proposed etiologies, risk factors, and biomarkers for the development of these disorders and for disease progression

Study Population:

240 patients with adult-onset progressive spasticity with a diagnosis of primary lateral sclerosis or related upper motor neuron disorder

Design:

Patients who have been referred by physicians for primary lateral sclerosis will undergo a screening evaluation at the first visit. The screening visit will include review of outside medical records, neurological examination, and diagnostic testing to determine possible causes of spasticity. Patients fulfilling the clinical criteria for primary lateral sclerosis by history or examination will be followed to determine the natural history of this disorder. Measures of motor and cognitive function will be made at baseline and follow-up visits to follow clinical progression. Magnetic resonance imaging will be carried out to determine if imaging changes occur over time. Blood samples may be collected for measurement of potential etiologies of PLS, including risk factor genes. Patients identified in this protocol who are eligible for other research protocols will be invited to participate in additional protocols.

Outcome Measures:

Clinical progression will be documented by measures of finger-tapping, timed gait, speech. The association between clinical progression and MRI measures will be assessed as a secondary outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 years of age or older
* Adult onset of progressive spasticity
* No family history of a similar disorder
* Able to provide consent or with a legally-authorized representative who can provide consent

EXCLUSION CRITERIA:

* History of stroke, cerebral palsy, traumatic brain injury or other known etiology of spasticity
* Non-neurological disorders producing muscle stiffness, such as fasciitis or rheumatological conditions
* Disorders in which pain limits the ability to move muscles, such as fibromyalgia or complex regional pain syndromes
* Profound weakness of voluntary movement
* Inability to travel to NIH
* Anticoagulation will be an exclusion for needle EMG studies
* Implanted devices or metal fragments in the brain or spinal cord will be an exclusion for MRI scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2001-05-01; Study Completion 2019-04-24

PRIMARY OUTCOMES:
The primary outcome of this protocol is to document the natural history of clinical progression in PLS, defined as the change in clinical measures of movement speed over time: finger tapping, timed gait, and time to read a standard passage.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Floeter, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Leclerc KM, Landry FJ. Benign nocturnal leg cramps. Current controversies over use of quinine. Postgrad Med. 1996 Feb;99(2):177-8, 181-4. PMID 8632965
- [Background] Bentley S. Exercise-induced muscle cramp. Proposed mechanisms and management. Sports Med. 1996 Jun;21(6):409-20. doi: 10.2165/00007256-199621060-00003. PMID 8784961
- [Background] Auger RG. AAEM minimonograph #44: diseases associated with excess motor unit activity. Muscle Nerve. 1994 Nov;17(11):1250-63. doi: 10.1002/mus.880171103. PMID 7935547
- [Derived] Clark MG, Smallwood Shoukry R, Huang CJ, Danielian LE, Bageac D, Floeter MK. Loss of functional connectivity is an early imaging marker in primary lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Nov;19(7-8):562-569. doi: 10.1080/21678421.2018.1517180. Epub 2018 Oct 9. PMID 30299161